CLINICAL TRIAL: NCT06976463
Title: Assessment of Parental Knowledge and Confidence in Providing First Aid for Choking and Infant Cardiopulmonary Resuscitation (CPR)
Brief Title: Parental Knowledge of First Aid for Choking and Cardiopulmonary Resuscitation in Infants Under One Year of Age
Status: Recruiting | Type: Observational
Sponsor: Andrzej Frycz Modrzewski Krakow University (Other)
Responsible Party: Principal Investigator, Renata Bakalarz, Principal Investigator, Andrzej Frycz Modrzewski Krakow University
Other Study IDs: KBKA/46/O/2024
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Choking in Infants; Cardiopulmonary Resuscitation (CPR); First Aid Training; Parental Knowledg
Keywords: Infant CPR, First Aid, Choking, Parental Knowledge, Emergency Response, Neonatal Resuscitation, First Aid Training
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- First Aid Knowledge Training Group (Pre-Post Evaluation): This group consists of parents of infants under one year of age participating in first aid training focused on cardiopulmonary resuscitation (CPR) and choking prevention. The aim is to assess parental knowledge and confidence in first aid techniques before and after the training. The training includes both theoretical and practical components, focusing on emergency response skills, proper CPR technique for infants, and choking management. The educational sessions are conducted in two formats: in-person workshops at selected hospitals and online via Zoom. Data collection will occur at two time points: before the training (baseline assessment) to evaluate initial knowledge and confidence levels, and after the training (follow-up assessment) to measure improvements. The training aims to increase parents' competence in handling emergency situations involving infants.

SUMMARY:
This study aims to assess the knowledge of parents regarding first aid for choking and cardiopulmonary resuscitation (CPR) in infants under one year of age. The primary objective is to evaluate how well parents understand emergency procedures and identify factors influencing their knowledge and confidence. The study will involve a combination of surveys and practical training sessions conducted both in-person and online.

DETAILED DESCRIPTION:
The study aims to evaluate the level of knowledge and self-confidence among parents regarding first aid procedures for choking and cardiopulmonary resuscitation (CPR) in infants under one year of age. The research will investigate the factors that influence parental knowledge, including previous first aid training, educational background, and prior experience in emergency situations.

The study will employ a mixed-methods approach, including both quantitative and qualitative data collection. Participants will complete structured surveys before and after training sessions to assess changes in knowledge and confidence levels. The primary training will be conducted through workshops at the Andrzej Frycz Modrzewski Krakow University and the Stefan Żeromski Specialist Hospital in Kraków. Additionally, online training will be offered via the Zoom platform to reach a broader audience.

The results will be statistically analyzed to identify key factors that improve parental first aid readiness. Findings are expected to contribute to the development of more effective educational strategies for parents, ultimately enhancing infant safety and emergency response skills.

ELIGIBILITY:
Inclusion Criteria:

* Parents or legal guardians of infants under 1 year of age.
* Adults aged 18 years and older.
* Individuals willing to participate in first aid training on choking prevention.
* Persons who provide informed consent for participation.

Exclusion Criteria:

* Lack of consent to participate in the study.
* Individuals under 18 years of age.
* Professionals in medical rescue or those with advanced first aid knowledge.
* Parents of children older than 1 year.
* Individuals unable to attend in-person or online training sessions.
* Health conditions that prevent participation in training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of parents and legal guardians of infants under one year of age. Participants include both mothers and fathers who are willing to participate in a first aid training program focused on choking prevention and management in infants. The training is designed to improve parental knowledge and skills in providing immediate first aid during choking incidents. Recruitment will be conducted through both in-person invitations at hospitals and online through social media platforms targeting parents and caregivers. Eligible participants must be at least 18 years old. Individuals with professional experience in medical rescue or advanced first aid knowledge will be excluded to maintain uniformity in the baseline knowledge of the study group. The study aims to enhance the ability of parents to respond effectively in emergency situations involving choking in infants.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in parental knowledge of first aid for choking in infants | Before training (baseline) and immediately after training (follow-up).
  The primary outcome measure of this study is the improvement in parental knowledge of first aid techniques for choking in infants. This will be assessed by comparing pre- and post-training scores obtained through a standardized questionnaire designed to evaluate the understanding of choking recognition, the correct application of first aid procedures (including back blows and chest thrusts), and the ability to assess the infant's condition. The questionnaire will multiple-choice questions, covering key aspects of infant choking management. The baseline assessment will take place before the training session, and the follow-up assessment will be conducted one week after the training. The primary objective is to quantify the increase in knowledge and practical understanding among parents after participating in a structured first aid training program. Data analysis will focus on changes in score distribution between the pre- and post-training assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- Stefan Żeromski Specialist Hospital in Kraków, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to confidentiality and privacy concerns. The collected data will be used exclusively for the purpose of the current study and will not be made available to other researchers.